CLINICAL TRIAL: NCT05232656
Title: Impact of an Epic-integrated Safety Dashboard and Interactive Pre-discharge Checklist on Post-discharge Adverse Events
Brief Title: PREventing Adverse Events Post-Discharge Through Proactive Identification, Multidisciplinary Communication, and Technology
Acronym: PREDICT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Crico (Other)
Responsible Party: Principal Investigator, Anuj K. Dalal, MD, Associated Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018P001137
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Transitions of Care; General Medicine; Discharge Checklist; Adverse Event

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention (No Intervention): Usual care on three general medicine units.
  Patients/caregivers do no have access to the discharge preparation checklist. Providers do not have access to the safety dashboard.
- Post-intervention (Experimental): Patients/caregivers have access to the pre-discharge preparation checklist. Providers have access to patient safety dashboard.
  Interventions: Behavioral: Pre-Discharge Checklist and Patient Safety Dashboard

INTERVENTIONS:
Behavioral: Pre-Discharge Checklist and Patient Safety Dashboard — Pre-discharge preparation checklist for patients to assess discharge readiness. Patient safety dashboard for clinicians to proactively identify at-risk patients.
  Arms: Post-intervention

SUMMARY:
The goal of this study is to expand the use of previously developed patient safety dashboards and patient-centered discharge checklists to three general medicine units in an affiliated community hospital. The safety dashboard and interactive pre-discharge checklist are cognitive aids for clinicians and patients, respectively, that serve to facilitate early detection of patients at risk for preventable harm, including suboptimal discharge preparation. The aims of this study are to:

1. Enhance the safety dashboard and interactive pre-discharge checklist to include "smart" notifications for hospital-based clinicians when patients are at high risk for adverse events or have identified specific concerns related to discharge based on their checklist responses.
2. Expand intervention to general medical units at our community hospital-affiliate, BWFH.
3. Evaluate impact on post-discharge AEs for patients discharged from BWFH who are at risk for preventable harm and hospital readmission.

DETAILED DESCRIPTION:
Our project proposes to address gaps in functionality of commercially available EHR systems through evaluation of novel, EHR-integrated HIT tools. We previously designed, developed, and implemented the patient safety dashboard and interactive pre-discharge checklist to engage clinicians and patients in systematically addressing safety threats in each of several domains. By integrating clinical data of several different types, these tools serve to reduce cognitive load and improve decision-making for clinicians. In this way, these tools represent a preventative intervention that mitigates risk in each domain by suggesting corrective action corresponding to institutional safety guidelines.

Studying the effectiveness of these tools on post-discharge outcomes will improve knowledge, technical capability, and clinical practice related to patient safety during transitions of care. Specifically, our project will advance scientific knowledge by quantifying the post-discharge impact of an intervention that changes clinical practice by enabling hospital-based clinicians to proactively institute corrective action for "at risk" patients who may require additional surveillance and supportive services during transitions. Also, we will establish the technical feasibility of spreading customized, third-party digital health applications that fill critical safety gaps in commercially available EHRs; expanding to a community hospital has clear implications for adoption and validation of this technology in different practice settings.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, >18 years of age, English-speaking
* Caregivers >18 years of age designated by patient or patient's healthcare proxy
* Two or more patient safety risk factors

Exclusion Criteria:

- Non-English speaking patients for whom we cannot identify an English-speaking healthcare proxy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Potential Post-Discharge Adverse Events | 24 months
  Potential post-discharge adverse events will be measured as the number of new or worsening symptoms or signs per patient

SECONDARY OUTCOMES:
Actual Post-Discharge Adverse Events | 24 months
  Actual post-discharge adverse events will be measured as the number of adverse events per patient
Preventable Post-Discharge Adverse Events | 24 months
  Actual post-discharge adverse events related to preventable harm will be measured as the number of post-discharge adverse events per patient related to a specific safety risk domain identified during index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Anuj K Dalal, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vasudevan A, Plombon S, Piniella N, Garber A, Malik M, O'Fallon E, Goyal A, Gershanik E, Kumar V, Fiskio J, Yoon C, Lipsitz SR, Schnipper JL, Dalal AK. Effect of digital tools to promote hospital quality and safety on adverse events after discharge. J Am Med Inform Assoc. 2024 Oct 1;31(10):2304-2314. doi: 10.1093/jamia/ocae176. PMID 39013194